CLINICAL TRIAL: NCT00638911
Title: PMS Assessing the Safety and Efficacy of Telmisartan in Patients With Mild-to-moderate Essential Hypertension
Brief Title: Using Telmisartan Alone or Combination of Telmisartan -HCTZ in the Treatment of Mild to Moderate Essential Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.465
Record Dates: First submitted 2008-03-06; First posted 2008-03-19 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with hypertention

SUMMARY:
The aim of this therapeutic observation is to demonstrate the efficacy and safety of telmisartan or telmisartan and HCTZ in the treatment of patients with mild-to-moderate essential hypertension under normal conditions of use after market launch.

DETAILED DESCRIPTION:
Study 502.465(NCT00638911) was planned and conducted as 6 independent substudies with varying country participation. One study database, a data management plan or a TSAP were not planned and do not exist which precludes baseline and outcome analyses.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients over the age of 18 years, with mild-to-moderate essential hypertension with values of mean morning seated diastolic BP more than 90 mmHg and less than 109 mmHg and or mean morning seated systolic BP more than 140 mmHg and less than 180 mmHg

1. newly diagnosed patients
2. patients failing to reach target blood pressure of less than 140 on 90 on their current antihypertensive treatment

Exclusion criteria:

1. Pre-menopausal women who do not use adequate contraception who are pregnant or nursing
2. Cholestasis and biliary obstructive disorders
3. Severe hepatic impairment
4. Severe renal impairment creatinine clearance less than 30 ml pro min
5. Refractory hypokalaemia hypercalcaemia
6. Known hypersensitivity to any component in the formulation of Micardis/Micardis Plus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 33247 (Actual)
Dates: Start 2004-09; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Primary Endpoints will be the change from baseline in mean systolic blood pressure. | 4-24 Weeks

SECONDARY OUTCOMES:
Secondary Endpoints are clinical control of the BP and response rate. | 4-24 Weeks
Other secondary Endpoints will be discontinuations and tolerability. | 4-24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim